CLINICAL TRIAL: NCT07137585
Title: Effects of RO7204239 on Insulin Sensitivity, Muscle Composition and Function in Participants Living With Type 2 Diabetes Mellitus and Overweight or Obesity: A Double-blind, Randomized, Placebo-controlled Study
Brief Title: A Study to Evaluate the Effect of RO7204239 on Insulin Sensitivity and Muscle Composition in Participants With Type 2 Diabetes Mellitus (T2DM) and Overweight or Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP45980; 2025-521401-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental): Participants will receive RO7204239 matching placebo, every 4 weeks (Q4W), as a subcutaneous (SC) injection for 24 weeks.
  Interventions: Drug: Placebo
- RO7204239 (Experimental): Participants will receive RO7204239, Q4W, as a SC injection for 24 weeks.
  Interventions: Drug: RO7204239

INTERVENTIONS:
Drug: Placebo — RO7204239 matching placebo will be administered as per the schedule specified in the treatment arm.
  Arms: Placebo
Drug: RO7204239 — RO7204239 will be administered as per the schedule specified in the treatment arm.
  Other Names: GYM329
  Arms: RO7204239

SUMMARY:
The main purpose of this study is to assess the effect of RO7204239 on insulin sensitivity versus placebo in participants with T2DM and obesity or overweight.

ELIGIBILITY:
Inclusion Criteria:

* Participants with T2DM for at least 6 months, treated with diet, exercise and/or metformin alone or in combination with either dipeptidyl peptidase 4 (DPP-4) inhibitor or sodium-glucose co-transporter 2 (SGLT2) at stable dose for the last 3 months prior to study entry and with a HbA1c between ≤ 6.5% and ≤ 10%
* Body mass index (BMI) within the range of 27.0 to 45.0 kilogram per meter square (kg/m2)
* Stable body weight for the 3 months prior to screening
* Participants on lipid-lowering or antihypertensive drugs must be on stable doses for at least 3 months

Exclusion Criteria:

* Type 1 diabetes mellitus (DM), known latent autoimmune diabetes in adults, or people with an episode of ketoacidosis or hyperosmolar state requiring hospitalisation in 6 months prior to screening
* Active proliferative diabetic retinopathy, diabetic maculopathy, or severe non-proliferative diabetic retinopathy requiring acute treatment
* Uncontrolled comorbid conditions commonly associated with diabetes (for example, hypertension, hyperlipidaemia)
* Severe hypoglycaemia within 6 months prior to screening visit
* Current autonomic neuropathy as evidenced by neuropathic urinary retention, resting tachycardia, orthostatic hypotension, or diabetic diarrhea
* Have evidence of a significant, uncontrolled endocrine abnormality (e.g., thyrotoxicosis and adrenal crises)
* Are currently taking a central nervous system stimulant (e.g., Ritalin-SR), with the exception of caffeinated beverage
* Have a known allergy, hypersensitivity, or intolerance to any component of the study treatment (i.e., RO7204239 / placebo) formulation
* Blood donation of more than 500 milliliters (mL) within the past 3 months or blood transfusion or severe blood loss within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-09-13 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in M-value in a Hyperinsulinemic Euglycemic Glucose Clamp (HEC) at Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Glucose Metabolism Assessed Using Fasting Glucose Test at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Glucose Metabolism Assessed Using Insulin Test at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Glucose Metabolism Assessed Using C-peptide Test at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Blood Lipid Profiles at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Body Weight at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Waist Circumference at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Waist to Height Ratio at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Total Lean Tissue Volume and Total Adipose Tissue Volume From Abdominal Magnetic Resonance Imaging (MRI) at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Muscle Volume From Thigh Muscle MRI at Weeks 12 and 24 | Baseline, Week 12, Week 24
Change From Baseline in Muscle Fat Infiltration From Thigh Muscle MRI at Weeks 12 and 24 | Baseline, Week 12, Week 24
Number of Participants With Adverse Events (AEs) | Up to Week 48
Number of Participants With Local and Systemic Injection Reactions | Up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No